CLINICAL TRIAL: NCT05265507
Title: Comparison of Anti-nausea and Vomiting Effect After Elective Surgery Undergoing General Anesthesia Between Glycopyrronium and Ondansetron: a Multi-center Study
Brief Title: Comparison of Postoperative Anti-nausea and Vomiting Effect Between Glycopyrronium and Ondansetron
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: Chongqing University Jiangjin Hospital (Unknown); Chongqing Medical University (Other); The People's Hospital of DAZU ，Chongqing (Unknown); Xiangya Hospital of Central South University (Other); West China Hospital (Other); The People's Hospital of Tongliang District， Chongqing city (Unknown); Chongqing Medical Center for Women and Children (Other); Dianjiang People's Hospital of Chongqing (Unknown); The Ninth People's Hospital of Chongqing (Unknown); The People's Hospital of Yubei District of Chongqing city (Unknown); Chongqing Yongchuan District People's Hospital (Unknown); The First People's Hospital Of Chongqing Liang Jiang New Area (Unknown); ChongGang General Hospital (Unknown); The People's Hospital of Nanchuan (Unknown); People's Hospital of Pengshui County (Unknown); Yunyang people's Hospital (Unknown); Chongqing Liangping District People's Hospital (Unknown); Jiulongpo People's Hospital of chongqing (Unknown); The People's Hospital of Qijiang District，Chongqing (Unknown); University-Town Hospital of Chongqing Medical University (Other); Chongqing Public Health Medical Center (Other); CHONGQING BANAN HOSPITAL OF TCM (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Glycopyrronium and ondansetron
Record Dates: First submitted 2022-02-23; First posted 2022-03-03 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Glycopyrrolate; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glycopyrronium (Experimental): Glycopyrronium (0.2mg) was intravenously given at the ending of the surgery.
  Interventions: Drug: Glycopyrronium
- Ondansetron (Active Comparator): Ondansetron (4mg) was intravenously given at the ending of the surgery.
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Glycopyrronium — Glycopyrronium (0.2mg) was intravenously given at the ending of the surgery.
  Arms: Glycopyrronium
Drug: Ondansetron — Glycopyrronium (4mg) was intravenously given at the ending of the surgery.
  Arms: Ondansetron

SUMMARY:
To compare the anti-nausea and vomiting effect between glycopyrronium and ondansetron for patients receiving elective surgery under general anesthesia. Based on this study the investigators intend to explore the feasibility of using glycopyrronium to prevent postoperative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists classification I-III
* Receive general anesthesia
* Voluntarily receive postoperative intravenous controlled analgesia

Exclusion Criteria:

* Puerpera or lactation women
* Allergy or existing contraindication to glycopyrronium and ondansetron
* Participate in other clinical drug trials within three months
* Can not follow with the study procedure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
incidence of postoperative nausea and vomiting | from the ending of surgery to 24 hours after surgery
  postoperative nausea and vomiting is recorded according to follow-up visits after surgery

SECONDARY OUTCOMES:
intensity of postoperative nausea | from the ending of surgery to 24 hours after surgery
  intensity of postoperative nausea is assessed using Numeric Rating Scale (0-10, 0 represents no uncomfortable felling, 10 represents tolerableness)
incidence of postoperative vomiting | from the ending of surgery to 24 hours after surgery
  postoperative vomiting is recorded according to follow-up visits after surgery
incidence of intervention requirement for nausea and vomiting | from the ending of surgery to 24 hours after surgery
  this event is recorded according to follow-up visits after surgery

OTHER OUTCOMES:
Postoperative pain intensity | from the ending of surgery to 24 hours after surgery
  Pain intensity is assessed by numerical rating scale (0-10, 0 represents painless; 10 represents intolerable pain)
Postoperative analgesic requirements | from the ending of surgery to 24 hours after surgery
  Analgesic requirements is assessed by recording the volume of patient controlled analgesia pump
degree of satisfaction | from the ending of surgery to 24 hours after surgery
  degree of satisfaction is assessed by patient using numerical rating scale (0-10, 0 represents unsatisfactory; 10 represents complete satisfaction)
adverse reaction related to glycopyrronium and ondansetron | from the ending of surgery to 24 hours after surgery
  adverse reaction is recorded according to follow-up visits after surgery

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — The Second Affiliated Hospital, Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data for this study is available from the sponsor on reasonable request through email.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within five years